CLINICAL TRIAL: NCT06302088
Title: Safety Integration Stakeholders: A Randomized Control Trial to Minimize Patient Fall Risk and Reduce Patient-assist Injuries Among Critical Access Hospital Staff
Brief Title: The Safety Integration Stakeholders (SAINTS) Program to Integrate Worker and Patient Safety in Oregon Rural Hospitals
Acronym: SAINTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Hurtado, ScD, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00026205
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Accidental Falls; Injuries
Keywords: Patient falls; patient-assist injuries; safety climate
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: All participating clinics will take part in baseline surveys of unit staff (n=240-360) and safety stakeholders will be identified. Following surveys, hospitals will be randomized to the control arm (n=3) or the intervention arm (n=3). Both groups will engage in key informant interviews on safety culture (n=30-60). Control group hospitals will continue standard operating procedures. Intervention group hospitals will engage in social network analysis of surveys, have peer leaders identified, and engage in safety leadership training and quality improvement cycles. All hospitals regardless of arm will take part in 6-and-12-month surveys and 24-month interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control Arm (No Intervention): Control Arm engages in baseline, 6-and-12-month surveys, as well as baseline interviews and 24-month interviews. They engage in standard operating procedures and do not take part in the intervention
- SAINTS program Intervention Arm (Experimental): Intervention arm engages in baseline, 6-and-12-month surveys, as well as baseline interviews and 24-month interviews. They engage in safety training programs and quality improvement cycles during the duration of the intervention.
  Interventions: Other: SAINTS program

INTERVENTIONS:
Other: SAINTS program — A brief descriptive name used to refer to the intervention(s) studied in each arm of the clinical study. A non-proprietary name of the intervention must be used, if available. If a non-proprietary name is not available, a brief descriptive name or identifier must be used.
  Arms: SAINTS program Intervention Arm

SUMMARY:
The safety integration stakeholders (saints) program to integrate worker and patient safety in Oregon rural hospitals. The rationale is that the saints program will positively impact outcomes by identifying and training peer leaders on strategies to optimize environmental, administrative, and educational components to become a saint and regularly collaborate with safety stakeholders/administrative leaders at each site through continuous improvement cycles (e.g. plan-do-study-act).

DETAILED DESCRIPTION:
SAINTs program will follow a semi-structured, block randomized control design along with a multi-method process evaluation to identify the extent to which the program was delivered as planned and if it led to the adoption of preventative measures. RCT measures will consist of pre/post survey data (at 6 months, 12 months and 24 months) hosted through REDCap and available via link. Additional secondary, de-identified data in aggregate (e.g. # of patient falls, # of worker compensation claims) will supplement survey data. Process evaluation will consist of implementation logs and interviews with key players (safety and quality officers, front-line peer leaders). The semi-structured design allows for customization among different rural healthcare sites that will have unique resources and needs, therefore requiring unique, tailored solutions. The combination of qualitative and quantitative. The SAINTS program will be implemented in four stages. 1) involvement of patient and worker safety stakeholders (e.g., Employee Health and Safety Officer, Quality Director, unit medical directors), 2) use of Social Network Analysis (SNA) to identify peer-recognized safety leaders; 3) training modules to stakeholders on safety leadership, and 4)in implementation of QI cycles to address barriers to safe patient handling and mobility (SPHM).

ELIGIBILITY:
Inclusion Criteria:

* Employed at participating sites (critical-access hospitals in rural Oregon)
* Patient-care workers (e.g. RNs, CNAs)

Exclusion Criteria:

* Non-clinical staff (e.g. clerical, janitorial)
* Non-unit staff (e.g. physical therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety participation | Baseline and 12-month follow up surveys
  Shared perceptions that worker safety is a priority at a hospital. We will use the safety compliance scale developed by Neal and Griffin. A six-item scale will be used to measure this self-reported construct, including three items for safety compliance (e.g., "I use the correct safety procedures for carrying out my job") and another three items for safety participation (e.g., "I voluntarily carry out activities that help to improve workplace safety"). Higher scores mean higher safety participation.

IPD SHARING:
Plan to Share IPD: No